CLINICAL TRIAL: NCT00001984
Title: Tolerance Induction Following Human Renal Transplantation Using Treatment With a Humanized Monoclonal Antibody Against CD52 (Campath-1H)
Brief Title: Effectiveness of the Investigational Drug Campath-1H in Preventing Rejection of Transplanted Kidneys
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000013; 00-DK-0013
Record Dates: First submitted 2000-01-26; First posted 2000-01-27 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Graft Rejection; Kidney Disease
Keywords: Immunosuppression; Tolerance; DSG; Alemtuzumab
MeSH Terms: conditions — Kidney Diseases | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab and DSG (Experimental): The recipients of live donor kidneys were treated perioperatively with alemtuzumab and DSG and followed postoperatively without maintenance immunosuppression.
  Interventions: Drug: Alemtuzumab and DSG

INTERVENTIONS:
Drug: Alemtuzumab and DSG — Alemtuzumab was administered intravenously at 0.3 mg/kg/dose over 3 hr. Patients received one dose on each of days -1,+1,+3 and +5 relative to transplantation (total dose 1.2 mg/kg). Methylprednisolone was given prior to each dose to limit the cytokine release: 500 mg prior to dose 1, 125 mg prior to dose 2, and 60 mg prior to doses 3 and 4. Deoxyspergualin was dosed as follows. The first two patients received 4 mg/kg as a loading dose on the day of transplant and 2.5 mg/kg daily for 13 additional days (14 days of treatment; 36.5 mg/kg total dose). The next three patients received the same dosing regimen but it was initiated on postoperative day 12 to coincide with the resurgence of monocytes on days 12- 25.

SUMMARY:
This protocol will test a humanized monoclonal antibody known as Campath-1H for its ability to induce a state of permanent allograft acceptance, or tolerance, when administered in combination with a brief course of the immunosuppressive drug deoxyspergualin (DSG) at the time of human renal allotransplantation. Campath-1H is specific for the common lymphocyte and monocyte antigen CD52. Its administration temporarily depletes mature lymphocytes and some monocytes without altering neutrophils or hematopoietic stem cells. Deoxyspergualin inhibits the NFkB pathway thus preventing monocyte and macrophage activation.

Recipients of living or cadaveric donor kidneys will be treated with one dose of Campath-1H prior to transplantation to insure that peripheral depletion is achieved at the time of graft reperfusion. Three subsequent doses of Campath-1H will be administered on the first, third and fifth days after the transplant to deplete passenger donor leukocytes and residual recipient cells that mobilize in response to the allograft. In addition, patients will be treated with DSG for 14 days beginning on the day prior to surgery. This trial expands on pilot studies at the NIH of 15 patients in which Campath was given alone at the time of transplantation. In those studies, excellent peripheral depletion occurred after just one dose of Campath though central depletion required additional dosing. This allowed for greatly reduced immunosuppression to be used to prevent rejection, but to date, all patients have required some immunosuppressive medication. It is hoped that the addition of DSG will eliminate the need for long-term immunosuppression.

Patients will be followed closely in the post transplant period. If patients experience rejection, they will be treated with methylprednisolone and have immunosuppression added using sirolimus as the predominant immunosuppressive agent. In the previous phase of this study without DSG, this maneuver has in all cases been successful in returning the allograft to normal function.

In addition to evaluating graft function following transplantation, this protocol will also characterize and evaluate the function of the immune system and the composition of the T cell repertoire following the administration of Campath-1H and DSG, and during immune system recovery after transplantation.

DETAILED DESCRIPTION:
This protocol will test a humanized monoclonal antibody known as Campath-1H for its ability to induce a state of permanent allograft acceptance, or tolerance, when administered in combination with a brief course of the immunosuppressive drug deoxyspergualin (DSG) at the time of human renal allotransplantation. Campath-1H is specific for the common lymphocyte and monocyte antigen CD52. Its administration temporarily depletes mature lymphocytes and some monocytes without altering neutrophils or hematopoietic stem cells. Deoxyspergualin inhibits the Rel-B/ NFkB pathway thus preventing monocyte and macrophage activation. Extensive preliminary data have been accumulated in humans using Campath-1H and its non-humanized predecessors. Additionally, data have been generated using a similar depleting scheme with and without DSG in non-human primates. Both the human and non-human primate data suggest that profound mature mononuclear cell depletion establishes a window of opportunity during which foreign tissue can be transplanted without the need for additional immunosuppression. Regulatory events occuring during mature cell repopulation in the presence of allografted tissue created a state in which the graft may not be rejected even in the absence of chronic immunosuppression.

Recipients of living or cadaveric donor kidneys will be treated with one dose of Campath-1H prior to transplantation to insure that peripheral depletion is achieved at the time of graft reperfusion. Three subsequent doses of Campath-1H will be administered on the first, third and fifth days after the transplant to deplete passenger donor leukocytes and residual recipient cells that mobilize in response to the allograft. In addition, patients will be treated with DSG 4mg/kg/d x 1 beginning on day 12 and then 2.5 mg/kg/d for an additional 13 days. This trial expands on pilot studies at the NIH of 17 patients in which Campath was dosed both prior to and after transplantation with and without DSG. In those studies, excellent peripheral depletion occured after just one dose of Campath though central depletion required additional dosing. Thus, the goal of pre-reperfusion depletion can be achieved with a single pre-operative dose but thorough depletion requires additional post-operative dosing. Lasting rejection-free survival was not realized without the addition of some, albeit reduced immunosuppression. This is thought to be due to residual post-operative monocytes that infiltrated the allograft causing modest reversible allograft dysfunction. The current dosing regimen with DSG is thus designed to accomplish both pre-operative depletion, and more thorough post operative elimination of donor and recipient cells mobilizing as a result of reperfusion, combined with therapy aimed at preventing the activation of monocytes that escape depletion. The timing of the DSG is meant to correspond with the peripheral repopulation of monocytes seen in previous patients.

Patients will be followed closely in the post transplant period for evidence of a detrimental immune response to the allograft. In the previous patients experiencing graft directed immunity the graft dysfunction was preceded by a rise in activated monocytes in the peripheral blood and augmented transcription of the cytokine Tumor Necrosis Factor-alpha (TNF-a) in the allograft. This syndrome has been resistant to treatment with the TNF-a sequestrant Infliximab and is now thought to require more comprehensive monocyte directed therapy. If patients progress and graft dysfunction occurs, patients will be treated with methylprednisolone and have immunosuppression added using sirolimus as the predominant immunosuppressive agent. This maneuver has in all cases been successful in returning the allograft to normal function. Sirolimus has been chosen since it does not act by interfering with specific T cell receptor function, and thus, provides immunosuppressive coverage during cell repopulation without interfering with the antigen specific T cell events important for tolerance induction. Non-human primate and human clinical data support both of these approaches.

In addition to evaluating graft and patient outcome following transplantation, this protocol will also characterize and evaluate the function of the immune system and the composition of the T cell repertoire following the administration of Campath-1H and DSG, and during immune system recovery after transplantation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney transplant performed at the Warren G. Magnuson Clinical Center.

Willingness and legal ability to give informed consent, or permission from a legal guardian.

Willingness to travel to the Clinical Center for protocol specific samples to be taken, or in some cases, the ability to send samples via overnight mail.

Availability of donor tissue for testing. This could include splenic or peripheral blood lymphocytes from a cadaveric donor or a willing living donor enrolled on the Clinic Center Living Donor Protocol who consents to periodic phlebotomy for peripheral blood lymphocyte isolation.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 2 months prior to enrollment. Specifically, candidates must not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, antilymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive.

Any condition that precludes serial follow-up.

Any active malignancy or any history of a hematogenous malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are appropriately treated prior to transplant.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol allograft biopsies.

Platelet count less than 100,000/mm(3).

Hemoglobin less than 9.0 mg/dl. Patients may be on erythropoietin therapy, but will not be placed on therapy solely to facilitate research sample acquisition.

Any known immunodeficiency syndrome.

HLA identical status with a living donor.

Any history of uncompensated cardiac insufficiency, major vascular disease, or symptomatic coronary artery disease.

Systemic or pulmonary edema.

Inability to be effectively dialyzed.

Chronic hypotension (SBP less than 100 mmHg).

Any condition that would likely increase the risk of protocol participation or confound the interpretation of the data.

CMV negative status receiving an organ from a known CMV positive donor.

EBV negative status receiving an organ from a known EBV positive donor.

Panel reactive antibody greater than 20% due to HLA antibodies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1999-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Santiago-Delpin EA. Trends in kidney transplantation in the United States. Transplant Proc. 1998 Sep;30(6):2867-8. doi: 10.1016/s0041-1345(98)00846-x. No abstract available. PMID 9745602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five patients aged 28-54 years scheduled to receive their first live-donor kidney transplant were enrolled after informed consent for study participation was obtained.
Pre-assignment Details: Patients were excluded if they were: HLA identical with their donor; on immunosuppression within 6 months of enrollment; or medically unsuitable for transplantation. Cytomegalovirus negative recipients of cytomegalovirus positive grafts were excluded.
Period: Overall Study
Arm/Group | Alemtuzumab and DSG
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 40 [28 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Relationship between Donor and Recepient [Number; unit: participants]
  Living related | 3
  Living unrelated | 2
Cause of end-stage renal disease [Number; unit: participants]
  Membranous glomerulonephritis | 1
  IgA nephropathy | 1
  Polycystic kidney disease | 1
  Medullary cystic disease | 1
  Obstructive uropathy | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Renal Allograft Rejection
Description: The renal allograft tolerance was evaluated clinically, by flow cytometry, and by protocol biopsies analyzed immunohistochemically and with real-time polymerase chain reaction.
Time Frame: from day 1 to 24 months post operation
Measure: Number; unit: participant
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
participant | 5

2. Primary Outcome: Rejection Day of Onset
Description: The day on which the rejection onsets.
Time Frame: From day 1 to 2 years post operation
Measure: Median (Full Range); unit: day
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
day | 28 [24 to 32]

3. Secondary Outcome: Creatinine Level at 6 Month Post Operation
Time Frame: 6 month post operation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
mg/dL | 1.5 (0.5)

4. Secondary Outcome: Creatinine Level at Year 1 Post Operation
Time Frame: 1 year post operation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
mg/dL | 1.4 (0.4)

5. Secondary Outcome: Creatinine at 2 Years
Description: Creatinine level of donor recepient at 2 years after transplantation
Time Frame: 2 years post operation
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
mg/dL | 1.7 (0.3)

6. Primary Outcome: Rise in Serum Creatineine Above Posttransplant Nadir
Time Frame: 24-32 days post operation
Measure: Median (Full Range); unit: parcentage rise in serum creatineine
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
parcentage rise in serum creatineine | 58 [20 to 530]

7. Secondary Outcome: Monocyte Count
Time Frame: 4 day post operation
Measure: Median (Full Range); unit: cells/mm3
Arm/Group | Alemtuzumab and DSG
Number analyzed (Participants) | 5
cells/mm3 | 527 [370 to 1600]

ADVERSE EVENTS:
Arm/Group | Alemtuzumab and DSG
Serious Adverse Events (participants affected / at risk) | 5/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab and DSG (N=5)
Allograft Rejection (Renal and urinary disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab and DSG (N=5)
postbiopsy hemodynamically significant renal arteriovenous fistula (Renal and urinary disorders) | 1 (1)
Grade II chronic allograft nepharopathy with proteinuria (Renal and urinary disorders) | 2 (2)
Grade II CAN at year 1 post operation (Renal and urinary disorders) | 1 (1)
OKT3 rescue requirement (Renal and urinary disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No